CLINICAL TRIAL: NCT05861934
Title: The Effect of Distant Reiki Application on Pain, Functional Status and Sleep Quality in Rheumatoid Arthritis Patients
Brief Title: The Effect of Distant Reiki Application on Pain, Functional Status and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Cemile KÜTMEÇ YILMAZ, Principal Investigator, Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022/14-02
Record Dates: First submitted 2023-03-24; First posted 2023-05-17 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distant reiki group (Experimental): To examine the effect of distant reiki application on pain, functional status and sleep quality in rheumatoid arthritis patients.
  Interventions: Behavioral: Distant reiki group
- Control group (No Intervention): Control group; routine care and treatment will be applied.

INTERVENTIONS:
Behavioral: Distant reiki group — ccording to Classical Usui Reiki, Reiki II. Remote Reiki will be practiced twice a week for 6 weeks by researchers who have completed the Phase 2 training. The time of remote reiki application will be planned by talking with the patient.
  Arms: Distant reiki group

SUMMARY:
Rheumatoid Arthritis (RA) is a chronic, multisystemic, progressive autoimmune disease characterized by joint destruction in synovial tissue, causing joint swelling, pain and morning stiffness. It is estimated to affect 0.1%-2% of the world's adult population and more women than men. RA limits individuals' work, social, and home lives and functional capacities. Patients commonly experience pain and accompanying sleep problems. Interventions for these problems and symptom management are important. In this regard, this study was planned to examine the effect of distant reiki application on pain, functional status and sleep quality in rheumatoid arthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Not having a communication problem,
* Receiving outpatient treatment from the clinic where the research was conducted,
* To have the physical and cognitive competence to answer the data collection forms,
* Not having received body-mind therapy (yoga, reiki, meditation, etc.) in the last six months,

Exclusion Criteria:

* individuals who have done reiki therapy before
* Being under 18 years old,
* Hearing and speaking problems that prevent communication,
* Participating in yoga, reiki, meditation practices in the last 6 months,
* Individuals with cognitive and severe psychiatric problems who cannot answer the survey questions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Distant Reiki application changes the level of pain in rheumatoid arthritis patients. | 6 weeks
  Pain level will be assessed using the Visual Analog Scale as a pre-test before starting the distant reiki application and 6 weeks later as a post-test. (Distant Reiki will be applied for 30 minutes twice a week for 6 weeks).
Distant Reiki application changes the functional status in rheumatoid arthritis patients. Health Assessment Survey will be used to evaluate the functional status of patients in rheumatic diseases. | 6 weeks
  Functional status will be assessed using the Health Assessment Survey as a pre-test and 6 weeks later as a post-test. (Distant Reiki will be applied for 30 minutes twice a week for 6 weeks).
Distant Reiki application changes sleep quality in rheumatoid arthritis patients. Sleep quality will be assessed using the Pittsburgh Sleep Quality Index. | 6 weeks
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index as a pre- test and 6 weeks later as a post-test test. (Distant Reiki will be applied for 30 minutes twice a week for 6 weeks).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Cemile KÜTMEÇ YILMAZ, Merkez, Aksaray
  - Aksaray University Health Science Faculty, Aksaray

IPD SHARING:
Plan to Share IPD: No